CLINICAL TRIAL: NCT02663986
Title: A School-Based Program to Improve Children's Organizational Skills
Brief Title: Organizational Skill Training (OST) in Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-02090
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Organization, Time Management, and Planning (OTMP)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — dolichyl-diphosphooligosaccharide - protein glycotransferase; Methods; Organizations; Time Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organizational Skills Training (OST) Intervention (Experimental): To improve children's organizational functioning, OST focuses on four key skills.
  * Tracking Assignments
  * Managing Materials
  * Time Management
  * Task Planning
  Interventions: Behavioral: Organizational Skills Training (OST) Intervention

INTERVENTIONS:
Behavioral: Organizational Skills Training (OST) Intervention
  Other Names: Organization, Time Management, and Planning (OTMP)

SUMMARY:
The primary aim of this project is to address the need for an effective school-based intervention for elementary school-aged students with Organization, Time Management, and Planning (OTMP) deficits by adapting an evidence-supported clinic-based intervention so that it can be implemented in school settings. Investigators are learning to adapt an individual, clinic based program (OST-C) for children diagnosed with Attention Deficit Hyperactive Disorder (ADHD) to children with OTMP problems. Investigators will be collecting data . To this end, investigators will be collecting data on implementation (such as feasibility and acceptability), program development (what changes to the individual OST-C program were made based on findings during this study) and limited outcome data (repeated measures collection and pre- and post-treatment collection on a small sample, no control group).

ELIGIBILITY:
Inclusion Criteria:

* Children will be recruited based on their parents' interest level in having them participate in a program to improve their organizational skills.
* Investigators will consider feedback from their 3rd to 5th grade general education or inclusion classroom teacher based on OTMP problems difficulties that interfere with functioning (difficulty in morning routine or end-of-day packing up routine, a high percentage of incomplete or missing assignments, messy desk or Seat Sack).
* Investigators will not use specific cutoffs on normed measures for determining eligibility based on these difficulties, as the intention is to develop a program that can be easily disseminated.
* Availability to attend twice-weekly sessions with the OTMP trainer either during the school day (during a time when they would not be pulled from academic content) or during after-school hours.

Exclusion Criteria:

* Children with Mental Retardation will not participate in the study, due to the difficulty they would likely have understanding the content of the sessions.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-02-01; Primary Completion 2016-06-28 (Actual); Study Completion 2016-06-28 (Actual)

PRIMARY OUTCOMES:
Change in scoring on Children's Organizational Skills Scale | 10 Weeks
Change in score on Organizational Skills Scale-Parent (COSS-P) | 10 Weeks
Change in score on Children's Organizational Skills Scale- (COSS-C) | 10 Weeks
Change in score on Organizational Skills Scale-Teacher (COSS-T) Versions COSS-P, COSS-C, and COSS-T | 10 Weeks
  be used to assess OTMP functioning at home and at school
Change in Homework Problem Checklist (HPCL) Score | 10 Weeks
  The HPCL (Anesko, Schoiock, Ramirez, & Levine, 1987) was designed to assess various aspects of homework performance. Parents are requested to rate each of 20 homework problems on a scale from 0 = never a problem to 3 = very often a problem
Change in score on Academic Progress Report (APR) | 10 Weeks
  The APR (Abikoff et al, 2013) assesses proficiency in six academic subjects relative to standard expectations (1=Well below standard expected at this time of year; 3=At standard; 5=Well above standard). The sum of ratings across the six academic subjects is the unit of analysis. Reliability is acceptable (coefficient alpha = .84), and this measure is sensitive to OST treatment effects (Abikoff et al., 2013).
Change in score on Consumer Satisfaction Questionnaire (CSQ) | 10 Weeks
  To assess satisfaction with treatment, and to serve as an index of treatment credibility, a consumer satisfaction questionnaire adapted from McMahon and Forehand (2003), will be completed by parents and teachers at post-treatment. Items (rated 1-7) tap overall satisfaction with treatment, perceived improvement of the child on the problems of concern to parent or teacher respectively, and evaluation of treatment providers.
Measures of Feasibility | 10 Weeks
  Investigators will gather feasibility data based on completed activities during the study. They will record information about treatment training, number of groups run, number of students per group, scheduling challenges, number of meetings/contacts OST-S trainers had with teachers and parents, materials support, or any other items related to implementing the program will be recorded for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Howard B Abikoff, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No